CLINICAL TRIAL: NCT06164847
Title: Effectiveness of the Adherence for Exercise Rehabilitation in Older People (AERO) Program to Improve Adherence in People with Osteoporosis in a German Context: a Randomized Parallel, Pilot Study
Brief Title: Effectiveness of the Adherence for Exercise Rehabilitation in Older People (AERO) Program in People with Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hochschule Osnabruck (Other)
Collaborators: LMU Klinikum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSOS/2023/1/1
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Osteoporosis; Osteopenia; Bone Loss
Keywords: exercise adherence; exercise program; osteoporosis; older adults
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two groups (HEP, PT+AERO and HEP, PT-standard care) will receive the protocol at the same time period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of the hypothesis of this study to decrease performance biases. The statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AERO Program (Experimental): Before their first physiotherapy appointment, patients will be asked to respond to four specific questions to guide the treatment (see link below).
  After this, they will receive usual physiotherapy care and a HEP for managing osteoporosis. The number of exercises given for the HEP should minimally be three to maximum six, performed at least three days per week for 12 weeks (time of the final assessment).
  After providing the HEP, patients in the intervention group are asked questions which explore their subjective abilities of the COM-B Model (capability, opportunity, or motivation) of undertaking the exercise program. Based on these answers and with the help of further discussions with the patient, the physiotherapist makes an assessment and decides which domains of the COM-B model might be useful to target. In the following 30 minutes PT-sessions, the therapist suggests one or more specific actions to enhance adherence. The participants must attend at least 4 out of 6 sessions.
  Interventions: Behavioral: AERO Program
- Standard care (Active Comparator): The control group will receive six PT sessions as "standard care". The first session is 60 minutes and the following sessions are 30 minutes. In regular clinical practice, "standard care" for people with osteoporosis includes measures such as home exercise programs, mobilizations, soft tissue techniques, or training with gym equipment. The HEP in the control group is based on the physical assessment of the physical therapist. The therapists in the control group do not have any restrictions for the exercises chosen. The participants must attend at least 4 out of 6 sessions of the control program.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: AERO Program — HEP, identification of barriers for exercise using the COM-B model. Interventions for these barriers: Review of HEP, review of method of delivery, cues, reminders, discussion of barriers and problem solving, motivational interviewing, decision balance sheets, behavioural contract, goal setting reviews, monitoring calls (detailed description in the link below).
  Arms: AERO Program
Other: Standard Care — home exercise programs, mobilisations, soft tissue techniques, or training with gym equipment
  Arms: Standard care

SUMMARY:
The goal of this pilot study is to investigate the effect of an evidence-based adherence promoting intervention on exercise adherence of patients with osteoporosis. For this reason, a randomized controlled pilot trial with an intervention period of three months will be conducted.

Question I:

To which extent does an adherence-promoting intervention (AERO) have an effect on adherence to long-term exercise programs in patients with osteoporosis compared to conventional standard care with home-based exercise therapy?

Objective II:

Does the AERO Intervention influence fall risk factors such as functional lower extremity strength and fear of falling compared to conventional standard care plus home-based exercise therapy in patients with osteoporosis? Patients will be randomized to two groups: an intervention and a control group. Both groups will receive instructions for a home exercise program (HEP) during six physical therapy (PT) sessions.

The intervention group will receive a HEP and additionally the so-called AERO (Adherence for Exercise Rehabilitation in Older people) intervention within 6 PT-Sessions. The AERO program is a feasible intervention for boosting the exercise adherence of older people. The AERO intervention is an evidence-based adherence promoting intervention approach to help patients adhere to an exercise program.

The control group will receive six PT sessions as "standard care". In regular clinical practice in Germany "standard care" for people with osteoporosis include measures such as home exercise programs, mobilisations, soft tissue techniques, or training with gym equipment. This will be delivered based on each PT clinical reasoning with no additional motivation for adherence to the exercise program.

DETAILED DESCRIPTION:
"Osteoporosis is a disease which causes the bones to become porous, weak and fragile. The result: a higher risk of broken bones, known as fragility fractures. Pain, fear of falling as well as reduced physical and social activity are also known complications that immensely impact the quality of life of patients with osteoporosis.

A common treatment goal in osteoporosis is the reduction of falls and fractures. Next to medication and dietary changes physical activity plays an important role in managing osteoporosis. The effectiveness of physical activity in people with osteoporosis has already been established. Strengthening exercises targeting the lower extremities have shown the largest effect for the bone mineral density (BMD) measured at the neck of the femur. These results are also enclosed in the German Osteoporosis Guideline: enhancing strength, coordination, and balance by promoting regular physical activity as part of the prevention and basic treatment plan for osteoporosis.

To achieve these goals, exercise needs to be executed thoroughly for a prolonged period of time and therefore treatment adherence to these exercise programs is crucial. Adherence itself is defined by the World Health Organization (WHO) as: ".... 'the extent to which a person's behavior corresponds with agreed recommendations from a healthcare provider." People with osteoporosis often have problems to adhere with any exercise program prescribed. About 50% of the participants of exercise programs quit these programs after six months. Rodrigues et al., analyzed 54 studies using exercises and reported adherence rates between 51% and 100%.

Multiple reasons, which are being referred to as barriers (e.g., lack of time, family priorities, monetary issues) are proposed as being linked to non-adherence. Therefore, measures that promote adherence towards these regimens are needed to ensure the long-term effects and benefits of exercise programs. It is crucial that patients conform to the recommendations made by the health care providers. The best exercise program is unsuccessful if it is not being followed.

Based on the literature and a previous review conducted by our team, only a few studies were found that looked at ways for improving adherence in individuals with osteoporosis. However, none of these studies investigated adherence as a primary outcome but only as a secondary outcome in regard to a specific exercise program.

One study identified by the authors through manual search was the Adherence for Exercise Rehabilitation in older people (AERO) intervention. Although not targeted to subjects with osteoporosis, this evidence-based intervention was created to enhance Adherence for Exercise Rehabilitation in older people. However, this program has only been implemented in United Kingdom using other populations. Thus, the main objective of this project will be to determine whether an adherence enhancing intervention (AERO intervention) would improve the exercise adherence of people with osteoporosis doing a home exercise program compared to conventional standard care using home-based exercise therapy in a German context.

To the knowledge of the authors this would be the first study which examines exercise adherence as primary outcome measure. Another advantage of the chosen design is that it is the first study design known by the authors targeting subjects with osteoporosis in which the control group does not receive an adherence-promoting intervention and therefore the effect of this measure can be derived. With this study design group differences and possible effects of the AERO-Intervention can be demonstrated more easily.

Question I:

To which extent does an adherence-promoting intervention (AERO) have an effect on adherence to long-term exercise programs in patients with osteoporosis compared to conventional standard care with home-based exercise therapy?

Question II:

Does the AERO Intervention influence fall risk factors such as functional lower extremity strength and fear of falling compared to conventional standard care plus home-based exercise therapy in patients with osteoporosis? The goal of this pilot study is to investigate the effect of an evidence-based adherence promoting intervention to the exercise adherence of osteoporosis patients. For this reason, a randomized controlled pilot trial with an intervention period of three months will be conducted.

The baseline assessment will be conducted before the randomization in the first physical therapy (PT) session. After completing baseline assessments, then the patient will be immediately randomized to each of the interventions. The intervention period starts in both groups with the first treatment and lasts three months.

The final assessment will be conducted 12 weeks after the first PT treatment, the appointment for the final assessment will be scheduled after 6 PT sessions. Patients will be randomly assigned into a control group and an intervention group using a computer program generated by an external party. In order to warrant allocation concealment, numbered, opaque, and sealed envelopes will be used.

To ensure that both patient groups are neutral about the study's objective, the patients are being told that both treatments are equally effective. Therefore, the patient is not biased beforehand knowing that he/she is in the intervention or the control group.

Group description:

The intervention group will receive a HEP and additionally the so-called AERO intervention within 6 PT-Sessions. The AERO program is a feasible intervention for boosting the exercise adherence of older people. The AERO intervention is an evidence-based adherence promoting intervention approach to help patients adhere to an exercise program.

The AERO intervention is theoretically underpinned by the Behavioural Change Wheel (BCW) with the COM-B Model in its center (see link below). The authors choose this intervention for their study because of the robust theoretical underpinning.

The AERO intervention consists of various parts. Before their first physiotherapy appointment, patients will be asked to respond to four specific questions in the waiting room to guide the treatment.

After this, they will receive a routine physiotherapy assessment and treatment which includes the instruction of a HEP in addition to usual care for managing osteoporosis. The therapist can use the answers from the aforementioned questions and any following discussion in developing the HEP.

The number of exercises given should minimally be three to maximum six and they should be performed at least three days per week. Besides this, the therapists should advise their patients to exercise regularly. Combined with the given home exercise program, the patient should be able to reach the recommended 150 minutes of the WHO. Nevertheless, for the purpose of this study and ensuring an accurate representation of adherence, we will collect information about adherence with their home exercise program (type of exercise, repetitions and sets). The additional activities will not be considered on this outcome.

After the assessment and hand-out of the home-exercise program, patients in the intervention group are asked to answer another set of questions which explores their subjective abilities of the COM-B Model (capability, opportunity or motivation) of undertaking the exercise program. Based on these answers and with the help of further discussions with the patient, the physiotherapist makes an assessment which domains of the COM-B model might be useful to target. In the following PT-sessions the therapist suggests one or more specific actions to enhance adherence. The participants have to attend at least 4 out of 6 sessions of the program to be considered compliant with the therapy; otherwise, they will be analyzed as not compliant.

The control group will receive six PT sessions as "standard care". In regular clinical practice "standard care" for people with osteoporosis include measures such as home exercise programs, mobilisations, soft tissue techniques, or training with gym equipment. The HEP in the control group is based on the physical assessment of the physical therapist and the individual problems of the patient. If a patient presents with, e.g., reduced mobility of the spine, a suitable exercise will be applied. The therapists in the control group do not have any restrictions for the exercises chosen, they just need to be able to be performed at home without any major equipment. The therapist is advised to tell the patient how often they must exercise throughout the week. The participants have to attend at least 4 out of 6 sessions of the control program to be considered compliant with the therapy; otherwise, they will be analyzed as not compliant.

Statistical Analysis:

The demographics of study participants will be described and will be presented in a tabular fashion (i.e., height, weight, BMI, age and sex) and separated by groups. Mean (SD), median (interquartile range), frequencies will be used to describe the population.

To investigate the first objective of this study, if adherence-promoting interventions (AERO) influence adherence to long-term exercise programs in patients with osteoporosis compared to conventional exercise therapy, two analyses will be performed. One analysis will include within group and the other will include between groups. Due to the small sample size, we anticipate that our data will not be normally distributed, and therefore we will conduct nonparametric tests to determine our p values. These analyses will be complemented by parametric tests to confirm results (when possible).

To determine differences before and after each individual treatment, we will conduct a Wilcoxon matched pairs test or a bootstrapped dependent t-test for the adherence scale. Calculation of the effect size for each group will be also performed. To determine differences between treatments, we will conduct a Mann-Whitney test or a bootstrapped independent t-test for the adherence scale. The alpha Level will be set to p=0.05 for all analyses. The same analysis will be conducted for secondary outcomes such as the 30s chair stand and the FES-I. The data of the diary will be analyzed with the Chi-Square Test.

To investigate the second objective, if the AERO intervention influences the fear of falling and increases the functional lower extremity strength, the author plans to analyze the data for differences between the baseline data and the data after the observation period within one group. Therefore, authors plan to analyze the 30s chair stand and the FES-I via Wilcoxon-Rank Test. For differences in the data between the two groups the authors plan to analyze the OEE-2 and the 30s chair stand via Mann Whitney U.

Alpha Level will be set to p=0.05. The beta level will be set to 0.2. Since there is not a gold standard measure for adherence there also is not a minimal clinical change (MCD) or minimal clinical important difference (MCID) which could tell the difference in exercise adherence. Therefore, the authors will be only able to report the group differences and if they are significant or not. Effect sizes will be calculated to enlighten the clinical significance of these findings.

The statistical analysis will be performed by the main researchers of this project under supervision. The data will be blinded and therefore the authors would not be biased. Both authors have taken several lectures of statistical analysis and will work in cooperation with their research supervisor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoporosis by a physician.
* able to speak and understand German.
* women or men Age ≥ 50 years old.
* able to make one repetition of the 30s sit-to-stand test.
* Ability to perform Physical Therapy (PT) sessions and perform exercises (time/schedule/monetary).
* Be referred to physiotherapy by a physician.

Exclusion Criteria

* cognitive impairment/ unable to follow instructions of the physiotherapist.
* secondary bone loss due to other disorders or medication in the last 5 years (e.g., cancer).
* conditions that would make participation in this study unsafe or would confound the results (e.g., renal failure, heart failure, cardiac diseases, pacemaker).
* current participation in other physio-individual therapy or part stationary, multimodal therapy programs at the same time.
* acute fractures (fracture within the last 6 weeks).
* Mini Cognitive Score of ≤ 3

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Exercise adherence | Baseline-3 months
  Exercise adherence will be measured via Outcome Expectations for Exercise Scale-2 and (OEE-2 scale) and via self-reported exercise diaries. The chosen outcome expectations for exercise scale 2 is a 13-item self report questionnaire to assess negative and positive exercise outcome expectations in older adults and is validated to the German language. Nine items rank positive expectations, and four items rank negative expectations. Each item can be rated from 1 (strongly disagree) to 5 (strongly agree). Low mean scores in the positive expectations part of the OEE-2 indicate positive expectations of exercise, high mean scores indicate negative expectations of exercise. High mean scores in the negative expectations part of the OEE-2 indicate positive expectations, low mean scores in the negative expectations part of the OEE-2 indicate low expectations of exercise. This measurement was included to investigate if the AERO intervention changes the expectations of the patient about exercise.

SECONDARY OUTCOMES:
Functional lower extremity strength | Baseline-3 months
  Functional lower extremity strength will be measured via a 30s chair stand test. The 30-Second Chair Test is administered using a folding chair without arms, with a seat height of 43.2 cm (Jones et al. 1999). The chair is placed against a wall to prevent it from moving. The participant is seated in the middle of the chair, back straight, feet approximately a shoulder width apart, and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest. If the patient uses his hands to complete a repetition, this repetition is counted as 0. The patient is encouraged to complete as many full stands as possible in 30 seconds. The patient is advised to sit between each repetition (Jones et al. 1999). This measurement was included to measure clinical improvements that could result from an improved exercise adherence in patients with osteoporosis.
Fear of falling | Baseline-3 months
  Will be measured by the Falls Efficacy Scale International (FES-I). The FES-I is a 16-item patient related outcome measure. The patient is asked to rate each activity on a four-point Likert scale. The patients rate their fall risk if they do certain activities, regardless of whether they actually perform it. Items are scored with 1 if the patients are not concerned at all about falling during this activity, the item is scored by 4 if the patient is very concerned about falling. Then the items are summed up to calculate a total score, which ranges between 16 and 64 points. The higher the score the greater the fear of falling.

OTHER OUTCOMES:
Other variables of interest | Demographics: baseline, Therapeutic alliance: 3 months
  Demographic variables such as age and gender will be used to characterize the sample. Therapeutic alliance (TA): the relationship between the patient and the physiotherapist during the treatment, although not an outcome per se is another factor that has an impact on exercise adherence. Therefore, the authors decided to include the working alliance subscale of the Pain Rehabilitation Expectations Scale (PRES) from Cheing et al. (Cheing et al., 2010) to be able to represent this influencing factor better. The authors included the working alliance subscale, which consists of 11 items. Each item can be rated by a 4 -4-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = agree, and 4 = strongly agree) (Cheing et al. 2010). The total score of this questionnaire will be considered in the analysis part of this study as an adjusting factor.

CONTACTS AND LOCATIONS:
Locations (1):
- LMU Klinikum Großhadern, Munich, Bavaria, Germany

REFERENCES:
- [Background] Cummings SR, Cosman F, Lewiecki EM, Schousboe JT, Bauer DC, Black DM, Brown TD, Cheung AM, Cody K, Cooper C, Diez-Perez A, Eastell R, Hadji P, Hosoi T, Jan De Beur S, Kagan R, Kiel DP, Reid IR, Solomon DH, Randall S. Goal-Directed Treatment for Osteoporosis: A Progress Report From the ASBMR-NOF Working Group on Goal-Directed Treatment for Osteoporosis. J Bone Miner Res. 2017 Jan;32(1):3-10. doi: 10.1002/jbmr.3039. Epub 2016 Dec 27. PMID 27864889
- [Background] Benedetti MG, Furlini G, Zati A, Letizia Mauro G. The Effectiveness of Physical Exercise on Bone Density in Osteoporotic Patients. Biomed Res Int. 2018 Dec 23;2018:4840531. doi: 10.1155/2018/4840531. eCollection 2018. PMID 30671455
- [Background] Jack K, McLean SM, Moffett JK, Gardiner E. Barriers to treatment adherence in physiotherapy outpatient clinics: a systematic review. Man Ther. 2010 Jun;15(3):220-8. doi: 10.1016/j.math.2009.12.004. Epub 2010 Feb 16. PMID 20163979
- [Background] Lachman ME, Lipsitz L, Lubben J, Castaneda-Sceppa C, Jette AM. When Adults Don't Exercise: Behavioral Strategies to Increase Physical Activity in Sedentary Middle-Aged and Older Adults. Innov Aging. 2018 Jan;2(1):igy007. doi: 10.1093/geroni/igy007. Epub 2018 Apr 5. PMID 30003146
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Rodrigues IB, Armstrong JJ, Adachi JD, MacDermid JC. Facilitators and barriers to exercise adherence in patients with osteopenia and osteoporosis: a systematic review. Osteoporos Int. 2017 Mar;28(3):735-745. doi: 10.1007/s00198-016-3793-2. Epub 2016 Oct 6. PMID 27714441
- [Background] Room J, Dawes H, Boulton M, Barker K. The AERO study: A feasibility randomised controlled trial of individually tailored exercise adherence strategies based on a brief behavioural assessment for older people with musculoskeletal conditions. Physiotherapy. 2023 Mar;118:88-96. doi: 10.1016/j.physio.2022.08.006. Epub 2022 Aug 30. PMID 36266133
- [Background] Room J, Hannink E, Dawes H, Barker K. What interventions are used to improve exercise adherence in older people and what behavioural techniques are they based on? A systematic review. BMJ Open. 2017 Dec 14;7(12):e019221. doi: 10.1136/bmjopen-2017-019221. PMID 29247111
- [Background] Pinelli E, Barone G, Marini S, Benvenuti F, Murphy MH, Julin M, Kemmler W, Von Stengel S, Di Paolo S, Dallolio L, Maietta Latessa P, Zinno R, Bragonzoni L. Effects of COVID-19 Lockdown on Adherence to Individual Home- or Gym-Based Exercise Training among Women with Postmenopausal Osteoporosis. Int J Environ Res Public Health. 2021 Mar 2;18(5):2441. doi: 10.3390/ijerph18052441. PMID 33801389
- [Background] Wocken, K. M. (2013): Exercise Adherence in Older Adults. In: The international journal of behavioral nutrition and physical activity.
- [Background] Strüder, H. K. (2016): Leichtathletik. Trainings- und Bewegungswissenschaft - Theorie und Praxis aller Disziplinen. Unter Mitarbeit von Jonath, U., & Scholz, K. Köln: Sportverlag Strauß.
- [Background] Dachverband Osteologie: DVO-Leitlinie Osteoporose - Kitteltaschenversion
- See also: Study about the Behaviour change wheel, Pre & Post Physiotherapy Questions of the Intervention Arm, Interventions based on the AERO Program for the Intervention Arm — https://drive.google.com/drive/folders/1a2ctvNLSBi_xwyX3sQe1f8qKdasvu2AC?usp=sharing